CLINICAL TRIAL: NCT00438347
Title: Influence of Fitness on Brain and Cognition
Status: Completed | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Arthur Kramer, Director, Beckman Institute, University of Illinois at Urbana-Champaign
Other Study IDs: IA0102; 5R37AG025667-02 (NIH)
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Aging; Cognitive Ability, General
Keywords: Mild Cognitive Impairment; cognition disorders; brain health; psychological aspect of aging; exercise; physical fitness
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group 1: Intervention Group- aerobic exercise
  Interventions: Behavioral: Aerobic Exercise
- group 2: Control Group- stretching and toning
  Interventions: Behavioral: Stretching and toning

INTERVENTIONS:
Behavioral: Aerobic Exercise — One hour per day three times a week for one year
  Groups: group 1
Behavioral: Stretching and toning — One hour per day three times a week for one year
  Groups: group 2

SUMMARY:
The purpose of this study is to examine the effect of aerobic fitness training on human cognition, brain structure, and brain function of older adults.

DETAILED DESCRIPTION:
Recent studies have shown the encouraging effects of fitness training on human cognition, and brain structure and function. Such effects are of great interest both for what may they tell us about the nature of cognitive and brain aging and also for their public health implications. This study will test the hypotheses that: 1) improvements in aerobic fitness of older adults will lead to improved performance on a variety of cognitive processes, and especially those processes that are supported by frontal regions of the brain; 2) improvements in cognitive processes due to enhanced aerobic fitness will be visible on fMRI scans, and will be similar to those of young adults; 3) improvements in aerobic fitness, over the course of a 1 year intervention, will result in increases in gray and white matter volume.

One hundred forty sedentary older adults will be recruited for this study. Participants will be randomized to an aerobic exercise intervention group, or to a stretching and toning control group. Aerobic exercise sessions will be conducted three times a week for one year, beginning at a light to moderate intensity level over the first two months and progressing to a moderate to high level for the remainder of the year. The control group will meet on the same basis as the intervention group, and will participate in an organized program of stretching, limbering, and toning for the whole body that is specially designed for individuals 60 years of age and older.

During this time, participants will exercise, keep a daily exercise log detailing distance walked (routes will be measured and mapped for participants), time spent in aerobic activity, degree of intensity (rating of perceived exertion), general level of affect during exercise, resting and exercise heart rates. Participants will participate in the MRI/fMRI, physiological (cardiorespiratory) and psychosocial testing prior to the beginning of the fitness training intervention, following 6 months of fitness training, and at the conclusion of the 1 year of fitness training.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 75 years of age (for Sedentary Older Adults)
* Sedentary Older Adults: no physical activity in last six months; Young Comparison Sample: Moderately active lifestyle
* Capable of performing exercise
* Personal physician's examination and consent to participate in testing and exercise or control intervention
* Successful completion of graded exercise test without evidence of cardiac abnormalities or responses
* Adequate performance on the Pfeiffer (1979) Mental Status measure - Corrected (near and far) vision 20/40 or better
* Right-handed
* Intention to remain in the local area over the study period

Exclusion Criteria:

* Sedentary Older Adults: self reported physical activity on regular basis (2 times or more per week) in last six months; Young Comparison Sample: sedentary or highly active/athletic lifestyle
* Any physical disability that prohibits mobility (walking), stretching etc.
* Depression score on GDS indicative of clinical depression
* Presence of any implanted devices such as cardiac pacemakers or autodefibrillators; neural pacemakers, aneurysm clips in the CNS; cochlear implants; metallic bodies in the eye or CNS; any form of wires or metal devices that concentrate radiofrequency fields
* Left-handed
* Individuals with chronic inflammation (e.g. severe arthritis, psoriasis, inflammatory bowel disease, asthma, polyneuropathies, Lupus)
* Intent to move or take an extended vacation (i.e. longer than 1 month during the study period)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults over 60
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2006-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Behavioral measures | baseline, 6 and 12 months

SECONDARY OUTCOMES:
fMRI | baseline, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Art Kramer, PhD, Principal Investigator — Beckman Institute, University of Illinois
Locations (2):
- United States (2):
  - Beckman Institute, University of Illinois, Champaign, Illinois
  - University of Illinois, Urbana, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colcombe SJ, Kramer AF, Erickson KI, Scalf P, McAuley E, Cohen NJ, Webb A, Jerome GJ, Marquez DX, Elavsky S. Cardiovascular fitness, cortical plasticity, and aging. Proc Natl Acad Sci U S A. 2004 Mar 2;101(9):3316-21. doi: 10.1073/pnas.0400266101. Epub 2004 Feb 20. PMID 14978288
- [Background] Barnes DE, Yaffe K, Satariano WA, Tager IB. A longitudinal study of cardiorespiratory fitness and cognitive function in healthy older adults. J Am Geriatr Soc. 2003 Apr;51(4):459-65. doi: 10.1046/j.1532-5415.2003.51153.x. PMID 12657064
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Colcombe SJ, Erickson KI, Raz N, Webb AG, Cohen NJ, McAuley E, Kramer AF. Aerobic fitness reduces brain tissue loss in aging humans. J Gerontol A Biol Sci Med Sci. 2003 Feb;58(2):176-80. doi: 10.1093/gerona/58.2.m176. PMID 12586857
- [Derived] Fanning J, Porter G, Awick EA, Ehlers DK, Roberts SA, Cooke G, Burzynska AZ, Voss MW, Kramer AF, McAuley E. Replacing sedentary time with sleep, light, or moderate-to-vigorous physical activity: effects on self-regulation and executive functioning. J Behav Med. 2017 Apr;40(2):332-342. doi: 10.1007/s10865-016-9788-9. Epub 2016 Sep 1. PMID 27586134
- [Derived] Nagamatsu LS, Weinstein AM, Erickson KI, Fanning J, Awick EA, Kramer AF, McAuley E. Exercise Mode Moderates the Relationship Between Mobility and Basal Ganglia Volume in Healthy Older Adults. J Am Geriatr Soc. 2016 Jan;64(1):102-8. doi: 10.1111/jgs.13882. PMID 26782858
- [Derived] Gothe NP, Fanning J, Awick E, Chung D, Wojcicki TR, Olson EA, Mullen SP, Voss M, Erickson KI, Kramer AF, McAuley E. Executive function processes predict mobility outcomes in older adults. J Am Geriatr Soc. 2014 Feb;62(2):285-90. doi: 10.1111/jgs.12654. Epub 2014 Jan 21. PMID 24521364
- [Derived] Mullen SP, Wojcicki TR, Mailey EL, Szabo AN, Gothe NP, Olson EA, Fanning J, Kramer A, McAuley E. A profile for predicting attrition from exercise in older adults. Prev Sci. 2013 Oct;14(5):489-96. doi: 10.1007/s11121-012-0325-y. PMID 23412942
- [Derived] Wojcicki TR, Szabo AN, White SM, Mailey EL, Kramer AF, McAuley E. The perceived importance of physical activity: associations with psychosocial and health-related outcomes. J Phys Act Health. 2013 Mar;10(3):343-9. doi: 10.1123/jpah.10.3.343. Epub 2012 Jun 14. PMID 22820124
- [Derived] Mullen SP, Olson EA, Phillips SM, Szabo AN, Wojcicki TR, Mailey EL, Gothe NP, Fanning JT, Kramer AF, McAuley E. Measuring enjoyment of physical activity in older adults: invariance of the physical activity enjoyment scale (paces) across groups and time. Int J Behav Nutr Phys Act. 2011 Sep 27;8:103. doi: 10.1186/1479-5868-8-103. PMID 21951520
- [Derived] McAuley E, Mullen SP, Szabo AN, White SM, Wojcicki TR, Mailey EL, Gothe NP, Olson EA, Voss M, Erickson K, Prakash R, Kramer AF. Self-regulatory processes and exercise adherence in older adults: executive function and self-efficacy effects. Am J Prev Med. 2011 Sep;41(3):284-90. doi: 10.1016/j.amepre.2011.04.014. PMID 21855742
- [Derived] Szabo AN, Mullen SP, White SM, Wojcicki TR, Mailey EL, Gothe N, Olson EA, Fanning J, Kramer AF, McAuley E. Longitudinal invariance and construct validity of the abbreviated late-life function and disability instrument in healthy older adults. Arch Phys Med Rehabil. 2011 May;92(5):785-91. doi: 10.1016/j.apmr.2010.12.033. Epub 2011 Apr 1. PMID 21458777